CLINICAL TRIAL: NCT00119067
Title: Anthrax Vaccine Adsorbed: Human Reactogenicity and Immunogenicity Trial to Address Change in Route of Administration and Dose Reduction
Brief Title: Anthrax Vaccine Clinical Trial to Assess Dose Reduction and Route Change
Acronym: AVRP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Baylor College of Medicine (Other); University of Alabama at Birmingham (Other); Emory University (Other); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDC-NCID-3344
Record Dates: First submitted 2005-07-06; First posted 2005-07-13 (Estimated); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: Anthrax; Vaccine; Immunogenicity; Reactogenicity
MeSH Terms: conditions — Anthrax | interventions — Anthrax Vaccines; Biothrax; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Anthrax Vaccine Adsorbed 8-SQ (Active Comparator): receive 8 injections of AVA injected SQ at the same points as the original licensure: 0m, 2weeks, 1m, 6m, 12m, 18m, and 2 boosters - 30m and 42m.
  Interventions: Biological: Anthrax Vaccine Adsorbed
- Anthrax Vaccine Adsorbed 8-IM (Experimental): receive 8 injections of AVA IM administered at 0m, 2weeks, 1m, 6m, 12m, 18m, and 2 boosters - 30m and 42m.
  Interventions: Biological: Anthrax Vaccine Adsorbed
- Anthrax Vaccine Adsorbed 7-IM (Experimental): receive 7 injections of AVA IM administered at 0m, 1m, 6m, 12m, 18m, and 2 boosters - 30m and 42m.
  Interventions: Biological: Anthrax Vaccine Adsorbed
- Anthrax Vaccine Adsorbed 5-IM (Experimental): receive 5 injections of AVA IM administered at 0m, 1m, 6m, and 2 boosters - 30m and 42m.
  Interventions: Biological: Anthrax Vaccine Adsorbed
- Anthrax Vaccine Adsorbed 4-IM (Experimental): receive 4 injections of AVA IM; months 0, 2, 6 and a booster at month 42
  Interventions: Biological: Anthrax Vaccine Adsorbed
- Saline placebo IM or SQ (Placebo Comparator): Saline injections to be administered either IM or SQ at 0m, 2weeks, 1m, 6m, 12m, 18m, and 2 boosters - 30m and 42m.
  Interventions: Biological: Saline injection

INTERVENTIONS:
Biological: Anthrax Vaccine Adsorbed
  Other Names: AVA; BioThrax
  Arms: Anthrax Vaccine Adsorbed 4-IM; Anthrax Vaccine Adsorbed 5-IM; Anthrax Vaccine Adsorbed 7-IM; Anthrax Vaccine Adsorbed 8-IM; Anthrax Vaccine Adsorbed 8-SQ
Biological: Saline injection
  Arms: Saline placebo IM or SQ

SUMMARY:
Anthrax Clinical Trial Objectives:

To assess whether:

* Anthrax vaccine (AVA or BioThrax, BioPort Corp. Lansing MI) administered by the intramuscular (IM) route elicits antibody responses that are not inferior (i.e., "non-inferior") to that achieved by the currently licensed schedule.
* BioThrax administered by the IM route and containing fewer numbers of doses elicits antibody responses that are not inferior (i.e., "non-inferior") to that achieved by the currently licensed schedule.
* Differences in reactogenicity exist between the IM and subcutaneous (SQ) administration of BioThrax.

Additionally for the final report we will assess whether:

* Occurrence of adverse events following AVA administration is influenced by selected risk factors.

DETAILED DESCRIPTION:
This study is a 43-month prospective, randomized, double-blind, placebo-controlled comparison of immunogenicity and reactogenicity elicited by BioThrax given by different routes of administration (SQ versus IM) and dosing regimens (as many as 8 doses versus as few as 4 doses). Sterile saline is used as the placebo where doses are dropped in regimens using AVA, and in the all-placebo study group.

This study is conducted among a total of 1564 healthy adult men and women (18 to 61 years of age) at five sites in the United States. Participants were randomized into one of 6 study groups with 260 participants per group. One group receives BioThrax given as currently licensed (SQ with 6 doses followed by annual boosters); another group is given placebo IM (130 participants) or SQ (130 participants) in the currently licensed dosing regimen. The four other groups receive BioThrax IM in modified dosing regimens; placebo is given when a dose of BioThrax is omitted from the licensed dosing regimen. There are a total of 25 required visits for this study, during which all participants receive an injection of vaccine or placebo (8 injections total), have a blood sample drawn (16 or 17 total), and have an in-clinic examination for adverse events (22 total).

Immunogenicity is assessed by assaying 16 serial blood samples obtained from all participants and a 17th sample from a subset of participants before vaccination and at other specified times. Total anti-protective antigen IgG antibody (anti-PA IgG) is quantified using a standardized and validated enzyme-linked immunosorbent assay (ELISA); the primary study endpoints are 4-fold rise in antibody titer and antibody concentration relative to the pre-vaccination titers or assay reactivity threshold. A subset of serum samples is also assayed in an in vitro toxin neutralization assay (TNA) to measure the functional activity of anti-BioThrax antibodies. The kinetics of the immune response to BioThrax are examined at 3 time points in the study and blood samples from a subset of participants will be further tested in correlates of protection and immunogenetics substudies. All adverse events (AEs), including vaccine reactogenicity, are actively monitored. While all AEs will be ascertained among study participants, several endpoints will be defined based on the likelihood of their occurrence and/or their clinical importance. Of primary interest is the occurrence of local AEs such as warmth, tenderness, itching, pain, arm motion limitation, erythema, induration, nodule, and bruise. Systemic AEs such as fever, fatigue, muscle ache, headache, temperature, and painful axillary adenopathy are also evaluated.

This study is expected to provide the basis for consideration of change in route of BioThrax administration from SQ to IM and reduction in number of vaccine doses required for primary and booster immunization.

There is an interim analysis of data collected through each participant's first 7 months of this study for consideration in changing the route of BioThrax administration from SQ to IM, and elimination of the 2 week vaccine priming dose.

At the end of the study, the Sponsor will present the entire results of the trial to FDA for consideration in elimination of additional doses from the licensed BioThrax schedule. At that time, the Sponsor will also supplement these data with results from parallel non-human primate challenge studies and additional research on immunologic correlates of protection.

ELIGIBILITY:
Inclusion Criteria:

Read/sign Informed Consent Document; Female or male, 18 to 61 years old (up to 62nd birthday); Females must agree to exercise adequate birth control from the time of the screening procedures to one month after the last vaccination; willingness/ability to return for all follow-up visits and blood collections for the duration of the study; ability to understand/comply with planned study procedures; agree to complete the Participant Diary (Appendix G) and to report concomitant medications and AEs during the study period; thave two intact upper arms with sufficient subcutaneous and intramuscular tissue in the deltoid regions for vaccine administration.Potential participants with a history of the following conditions remain eligible for study enrollment: gestational diabetes; treated, controlled, uncomplicated hypertension; treated hypo- or hyperthyroidism; cured nonmetastatic cancer; disease-free for 5 years (excluding hematologic malignancies); localized skin cancer, resected (including squamous cell and basal cell carcinomas, participants with a history of melanoma must be disease-free for 5 years); exercise-induced bronchospasm; mild asthma: use of inhalers only for control of symptoms is acceptable (Persons who have required hospitalization for asthma within the previous 2 years or those who require chronic or frequent oral/parenteral steroids will not be eligible; use of low to medium doses of inhaled steroids; history of coronary artery disease, asymptomatic (NYHA Function Class I), on a stable medical regimen. Persons meeting these criteria must be at least 2 years post-myocardial infarction, cardiac bypass surgery, and/or percutaneous coronary intervention (e.g., angioplasty, stent placement, etc) in order to qualify. Persons with a history of cardiac disease must be under the care of a physician.

Exclusion Criteria:

Prior history of anthrax or immunization against anthrax; Known allergy to aluminum hydroxide, formaldehyde, benzethonium chloride, or latex; Pregnant/plans to become pregnant for duration of study/does not agree to use adequate birth control from the time of screening procedures to one month after last vaccination; Used cytotoxic therapy in previous 5 years; Cardiovascular disease with significant likelihood of progression over 5 years; Moderate to severe asthma, chronic obstructive pulmonary disease, other significant pulmonary disease; using high doses of inhaled steroids; Clinically recognized hepatic or renal insufficiency; Inflammatory, vasculitic, or rheumatic disease including systemic lupus erythematosis, polymyalgia rheumatica and rheumatoid arthritis, scleroderma; Known HIV, hepatitis B or hepatitis C infection; Other conditions known to produce or be associated with immune suppression; Neuropathy or other evolving neurologic condition; Unstable/moderate to severe mental illness; Ongoing drug abuse/dependence (including alcohol); Seizure disorder; Active malignancy or history of metastatic or hematologic malignancy; current diabetes; Anyone who plans to receive within 60 days of study entry: cytotoxic therapy, experimental products, a live vaccine outside this trial, immunosuppressive therapy, parenteral immunoglobulin or blood products; Anyone who plans to receive an inactivated vaccine outside this trial within 42 days after study entry;: experimental products, a live vaccine outside this trial, immunosuppressive therapy; Anyone who received an inactivated vaccine outside this trial within 14 days prior to study entry, parenteral immunoglobulin or blood products within three months of study. In addition to conditions listed above, temporary exclusion would result from moderate or severe illness and/or oral temperature >100.4˚F within 3 days of injection or chronic condition that, in opinion of investigator, would render injection unsafe or would interfere with evaluations.

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1564 (Actual)
Dates: Start 2002-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wright, DVM, Principal Investigator — Centers for Disease Control and Prevention
Locations (5):
- United States (5):
  - University of Alabama, Birmingham (UAB), Birmingham, Alabama
  - Emory, Atlanta, Georgia
  - Walter Reed Army Institute for Research (WRAIR), Silver Spring, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Baylor, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marano N, Plikaytis BD, Martin SW, Rose C, Semenova VA, Martin SK, Freeman AE, Li H, Mulligan MJ, Parker SD, Babcock J, Keitel W, El Sahly H, Poland GA, Jacobson RM, Keyserling HL, Soroka SD, Fox SP, Stamper JL, McNeil MM, Perkins BA, Messonnier N, Quinn CP; Anthrax Vaccine Research Program Working Group. Effects of a reduced dose schedule and intramuscular administration of anthrax vaccine adsorbed on immunogenicity and safety at 7 months: a randomized trial. JAMA. 2008 Oct 1;300(13):1532-43. doi: 10.1001/jama.300.13.1532. PMID 18827210
- [Result] Wright JG, Plikaytis BD, Rose CE, Parker SD, Babcock J, Keitel W, El Sahly H, Poland GA, Jacobson RM, Keyserling HL, Semenova VA, Li H, Schiffer J, Dababneh H, Martin SK, Martin SW, Marano N, Messonnier NE, Quinn CP. Effect of reduced dose schedules and intramuscular injection of anthrax vaccine adsorbed on immunological response and safety profile: a randomized trial. Vaccine. 2014 Feb 12;32(8):1019-28. doi: 10.1016/j.vaccine.2013.10.039. Epub 2013 Dec 25. PMID 24373307
- [Derived] Quinn CP, Sabourin CL, Schiffer JM, Niemuth NA, Semenova VA, Li H, Rudge TL, Brys AM, Mittler RS, Ibegbu CC, Wrammert J, Ahmed R, Parker SD, Babcock J, Keitel W, Poland GA, Keyserling HL, El Sahly H, Jacobson RM, Marano N, Plikaytis BD, Wright JG. Humoral and Cell-Mediated Immune Responses to Alternate Booster Schedules of Anthrax Vaccine Adsorbed in Humans. Clin Vaccine Immunol. 2016 Apr 4;23(4):326-38. doi: 10.1128/CVI.00696-15. Print 2016 Apr. PMID 26865594
- [Derived] Falola MI, Wiener HW, Wineinger NE, Cutter GR, Kimberly RP, Edberg JC, Arnett DK, Kaslow RA, Tang J, Shrestha S. Genomic copy number variants: evidence for association with antibody response to anthrax vaccine adsorbed. PLoS One. 2013 May 31;8(5):e64813. doi: 10.1371/journal.pone.0064813. Print 2013. PMID 23741398
- [Derived] Pajewski NM, Parker SD, Poland GA, Ovsyannikova IG, Song W, Zhang K, McKinney BA, Pankratz VS, Edberg JC, Kimberly RP, Jacobson RM, Tang J, Kaslow RA. The role of HLA-DR-DQ haplotypes in variable antibody responses to anthrax vaccine adsorbed. Genes Immun. 2011 Sep;12(6):457-65. doi: 10.1038/gene.2011.15. Epub 2011 Mar 3. PMID 21368772

RESULTS

PARTICIPANT FLOW:
Groups:
- Anthrax Vaccine Adsorbed 8-SQ: receive 8 injections of AVA injected SQ at the same points as the original licensure: 0m, 2weeks, 1m, 6m, 12m, 18m, and 2 boosters - 30m and 42m.
  Anthrax Vaccine Adsorbed
- Anthrax Vaccine Adsorbed 8-IM: receive 8 injections of AVA IM administered at 0m, 2weeks, 1m, 6m, 12m, 18m, and 2 boosters - 30m and 42m.
  Anthrax Vaccine Adsorbed
- Anthrax Vaccine Adsorbed 7-IM: receive 7 injections of AVA IM administered at 0m, 1m, 6m, 12m, 18m, and 2 boosters - 30m and 42m.
  Anthrax Vaccine Adsorbed
- Anthrax Vaccine Adsorbed 5-IM: receive 5 injections of AVA IM administered at 0m, 1m, 6m, and 2 boosters - 30m and 42m.
  Anthrax Vaccine Adsorbed
- Anthrax Vaccine Adsorbed 4-IM: receive 4 injections of AVA IM; months 0, 2, 6 and a booster at month 42
  Anthrax Vaccine Adsorbed
Period: Overall Study
Arm/Group | Anthrax Vaccine Adsorbed 8-SQ | Anthrax Vaccine Adsorbed 8-IM | Anthrax Vaccine Adsorbed 7-IM | Anthrax Vaccine Adsorbed 5-IM | Anthrax Vaccine Adsorbed 4-IM | Saline Placebo IM or SQ
Started | 260 (One person consented and enrolled, then withdrew prior to first vaccination.) | 262 | 256 | 258 | 268 | 260
Completed | 148 | 157 | 146 | 144 | 158 | 144
Not Completed | 112 | 105 | 110 | 114 | 110 | 116

BASELINE CHARACTERISTICS:
Population: mean study group size was 261 (range 260-268); proportions of men 48.8% to women 51.2% was not statistically different across groups or time points; mean age was 39 years; Whites accounted for 74%, Blacks for 21%, and "other" for 5% of participants; less than 5% of study population was Hispanic
Groups:
- Anthrax Vaccine Adsorbed 8-SQ: receive 8 injections of Anthrax Vaccine Adsorbed injected SQ at the same points as the original licensure: 0m, 2weeks, 1m, 6m, 12m, 18m, and 2 boosters - 30m and 42m.
- Anthrax Vaccine Adsorbed 8-IM: receive 8 injections of Anthrax Vaccine Adsorbed IM administered at 0m, 2weeks, 1m, 6m, 12m, 18m, and 2 boosters - 30m and 42m.
- Anthrax Vaccine Adsorbed 7-IM: receive 7 injections of Anthrax Vaccine Adsorbed IM administered at 0m, 1m, 6m, 12m, 18m, and 2 boosters - 30m and 42m.
- Anthrax Vaccine Adsorbed 5-IM: receive 5 injections of Anthrax Vaccine Adsorbed IM administered at 0m, 1m, 6m, and 2 boosters - 30m and 42m.
- Anthrax Vaccine Adsorbed 4-IM: receive 4 injections of Anthrax Vaccine Adsorbed IM; months 0, 2, 6 and a booster at month 42
- Total: Total of all reporting groups
Arm/Group | Anthrax Vaccine Adsorbed 8-SQ | Anthrax Vaccine Adsorbed 8-IM | Anthrax Vaccine Adsorbed 7-IM | Anthrax Vaccine Adsorbed 5-IM | Anthrax Vaccine Adsorbed 4-IM | Saline Placebo IM or SQ | Total
Number analyzed (Participants) | 259 | 262 | 256 | 258 | 268 | 260 | 1563
Age, Customized [Number; unit: participants]
  Age <30 | 77 | 63 | 75 | 77 | 72 | 75 | 439
  Age 30-39 | 42 | 57 | 77 | 65 | 60 | 60 | 361
  Age 40-49 | 91 | 87 | 54 | 64 | 91 | 73 | 460
  Age 50-61 | 49 | 55 | 50 | 52 | 45 | 52 | 303
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 135 | 132 | 131 | 136 | 132 | 800
  Male | 125 | 127 | 124 | 127 | 132 | 128 | 763
Race/Ethnicity, Customized [Number; unit: participants]
  Race: White | 199 | 197 | 194 | 183 | 201 | 185 | 1159
  Race: Black | 47 | 48 | 49 | 62 | 59 | 59 | 324
  Race: Other | 13 | 17 | 13 | 13 | 8 | 16 | 80
  Ethnicity:Non-Hispanic | 246 | 250 | 247 | 243 | 256 | 251 | 1493
  Ethnicity: Hispanic | 13 | 12 | 9 | 15 | 12 | 9 | 70

OUTCOME MEASURES:

1. Primary Outcome: Local AEs
Description: warmth, tenderness, itching, pain, arm motion limitation, erythema, induration, nodule, and bruise.
  The number of injections analyzable varies for each event based on the presence or absence of reported data.
Time Frame: 4 weeks after each injection
Population: There are missing data
Measure: Number; unit: injections
Units Other Than Participants: Number of doses received
Groups:
- SQ Females: female participants receiving SQ AVA injection
- IM Female: female participants receiving IM AVA injection
- SQ Males: male participants receiving SQ AVA injection
- IM Male: male participants receiving IM AVA injection
Arm/Group | SQ Females | IM Female | SQ Males | IM Male
Number analyzed (Participants) | 134 | 534 | 125 | 510
Number analyzed (Number of doses received) | 958 | 2806 | 835 | 2584
injections
  Warmth: number analyzed (Number of doses received) | 952 | 2772 | 827 | 2556
  Warmth | 500 | 344 | 186 | 189
  Tenderness: number analyzed (Number of doses received) | 952 | 2806 | 832 | 2584
  Tenderness | 667 | 1398 | 410 | 1075
  Itching: number analyzed (Number of doses received) | 946 | 2762 | 824 | 2551
  Itching | 247 | 160 | 80 | 77
  Pain: number analyzed (Number of doses received) | 942 | 2780 | 826 | 2561
  Pain | 201 | 569 | 96 | 341
  Arm Motion Limitation: number analyzed (Number of doses received) | 943 | 2771 | 822 | 2558
  Arm Motion Limitation | 94 | 434 | 50 | 218
  Erythema: number analyzed (Number of doses received) | 958 | 2791 | 835 | 2565
  Erythema | 723 | 952 | 399 | 603
  Induration: number analyzed (Number of doses received) | 946 | 2772 | 830 | 2555
  Induration | 411 | 386 | 195 | 245
  Edema: number analyzed (Number of doses received) | 948 | 2772 | 827 | 2558
  Edema | 345 | 528 | 225 | 354
  Nodules: number analyzed (Number of doses received) | 947 | 2762 | 825 | 2554
  Nodules | 409 | 161 | 133 | 98
  Bruise: number analyzed (Number of doses received) | 942 | 2764 | 822 | 2552
  Bruise | 69 | 150 | 65 | 32

2. Primary Outcome: Systemic AEs
Description: Fatigue, Muscle Ache, Headache, Fever, Tender Axillary Lymphnode The number of injections analyzable varies for each event based on the presence or absence of reported data.
Time Frame: 4 weeks after each injection
Population: We analyzed by number of doses received. There might be missing data; people dropped out as time went on
Measure: Number; unit: injections
Units Other Than Participants: Number of doses received
Arm/Group | SQ Females | IM Female | SQ Males | IM Male
Number analyzed (Participants) | 134 | 534 | 125 | 510
Number analyzed (Number of doses received) | 958 | 2806 | 835 | 2584
injections
  Fatigue: number analyzed (Number of doses received) | 942 | 2768 | 825 | 2564
  Fatigue | 118 | 278 | 69 | 182
  Muscle Ache: number analyzed (Number of doses received) | 942 | 2769 | 825 | 2558
  Muscle Ache | 57 | 226 | 36 | 132
  Headache: number analyzed (Number of doses received) | 942 | 2767 | 823 | 2559
  Headache | 90 | 219 | 39 | 105
  Fever: number analyzed (Number of doses received) | 937 | 2745 | 822 | 2546
  Fever | 0 | 0 | 0 | 1
  Tender Axillary Adenopathy: number analyzed (Number of doses received) | 939 | 2762 | 823 | 2553
  Tender Axillary Adenopathy | 10 | 17 | 3 | 8

3. Primary Outcome: Anti-protective Antigen IgG Geometric Mean Concentration
Description: Geometric mean of the Anti-PA IgG Concentration measured in μg/mL. The lower limit of quantification (LLOQ) is 3.7, results below the LLOQ have been replaced by 1/2 LLOQ (1.85) before taking the geometric mean.
Time Frame: 4 weeks after the m1, m6 and m42 injections
Measure: Geometric Mean (95% Confidence Interval); unit: μg/ml
Groups:
- Anthrax Vaccine Adsorbed 4-IM: receive 4 injections of AVA IM; 0m, 1m, 6m and a booster at 42m.
  Anthrax Vaccine Adsorbed
- Anthrax Vaccine Adsorbed 754-IM: The 7-IM, 5-IM, and 4-IM arms received the same 0, 1, 6 month primary series schedule, so were combined for analysis at months 2 and 7. Analysis at month 43 was done separately since the schedules differed at that time. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results.
Arm/Group | Anthrax Vaccine Adsorbed 8-SQ | Anthrax Vaccine Adsorbed 8-IM | Anthrax Vaccine Adsorbed 7-IM | Anthrax Vaccine Adsorbed 5-IM | Anthrax Vaccine Adsorbed 4-IM | Anthrax Vaccine Adsorbed 754-IM | Saline Placebo IM or SQ
Number analyzed (Participants) | 235 | 234 | 139 | 141 | 157 | 698 | 243
μg/ml
  Month 2 | 94.3 [82.1 to 108.3] | 84.5 [73.7 to 96.8] | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | 46.4 [42.2 to 51.0] | 1.9 [1.9 to 2.0]
  Month 7 | 201.1 [174.7 to 231.6] | 232.6 [202.4 to 267.3] | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | 206.9 [187.1 to 227.0] | 1.9 [1.9 to 2.0]
  Month 43 | 216.8 [185.8 to 253.1] | 320.5 [276.0 to 372.1] | 254.8 [222.0 to 292.4] | 310.0 [270.5 to 355.3] | 433.2 [379.6 to 494.4] | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | 1.9 [1.8 to 1.9]

4. Secondary Outcome: TNA ED50 Titer
Description: Geometric mean of the ED50. The ED50 is the reciprocal of the dilution at which patient serum neutralizes 50% of a dose of anthrax lethal toxin (ED50). The lower limit of quantification (LLOQ) for this assay is 36, results below the LLOQ have been replaced with 1/2 LLOQ (18) before taking the geometric mean. Note that this secondary endpoint was only performed on ~47% of the participants.
Time Frame: 4 weeks after the m1, m6 and m42 injections
Measure: Geometric Mean (95% Confidence Interval); unit: ED50 Dilutional Titer
Arm/Group | Anthrax Vaccine Adsorbed 8-SQ | Anthrax Vaccine Adsorbed 8-IM | Anthrax Vaccine Adsorbed 7-IM | Anthrax Vaccine Adsorbed 5-IM | Anthrax Vaccine Adsorbed 4-IM | Anthrax Vaccine Adsorbed 754-IM | Saline Placebo IM or SQ
Number analyzed (Participants) | 112 | 103 | 56 | 67 | 66 | 315 | 124
ED50 Dilutional Titer
  Month 2 | 229.1 [190.9 to 274.9] | 240.8 [196.5 to 295.2] | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | 165.5 [146.2 to 187.4] | 18.0 [18.0 to 18.0]
  Month 7 | 1281.1 [1073.9 to 1528.3] | 1630.0 [1354.3 to 1961.7] | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | 1423.9 [1253.1 to 1617.9] | 18.1 [17.9 to 18.4]
  Month 43 | 1015.0 [827.8 to 1244.4] | 1540.3 [1274.6 to 1861.4] | 1451.0 [1139.5 to 1847.7] | 1876.2 [1603.1 to 2195.9] | 2825.9 [2175.2 to 3671.3] | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | 18.0 [18.0 to 18.0]

5. Primary Outcome: Anti-protective Antigen IgG Geometric Mean Titer
Description: Geometric mean of the Dilutional Titer. The Dilutional Titer is the reciprocal of the dilution at which the anti-PA IgG response reaches a threshold. The lower limit of quantification (LLOQ) is 58, results below the LLOQ have been replaced by 1/2 LLOQ (29) before taking the geometric mean.
Time Frame: 4 weeks after the m1, m6 and m42 injections
Measure: Geometric Mean (95% Confidence Interval); unit: Dilutional Titer
Arm/Group | Anthrax Vaccine Adsorbed 8-SQ | Anthrax Vaccine Adsorbed 8-IM | Anthrax Vaccine Adsorbed 7-IM | Anthrax Vaccine Adsorbed 5-IM | Anthrax Vaccine Adsorbed 4-IM | Anthrax Vaccine Adsorbed 754-IM | Saline Placebo IM or SQ
Number analyzed (Participants) | 235 | 234 | 139 | 141 | 157 | 698 | 243
Dilutional Titer
  Month 2 | 1048.5 [913.1 to 1204.1] | 934.8 [815.6 to 1071.3] | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | 514.6 [468.1 to 565.7] | 29.7 [28.7 to 30.6]
  Month 7 | 2211.9 [1921.8 to 2545.9] | 2545.6 [2215.1 to 2925.1] | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | 2257.0 [2050.1 to 2484.9] | 29.7 [28.7 to 30.8]
  Month 43 | 2282.4 [1955.8 to 2663.5] | 3425.4 [2950.4 to 3976.9] | 2760.4 [2404.7 to 3168.6] | 3286.4 [2866.5 to 3767.8] | 4683.8 [4103.0 to 5346.8] | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | 29.0 [29.0 to 29.0]

6. Primary Outcome: 4-fold Rise in Anti-protective Antigen IgG Titer Response
Description: Percent of participants who achieved a 4-fold or greater rise in anti-PA IgG Titer relative to the pre-vaccination level at month 0. The Dilutional Titer is the reciprocal of the dilution at which the anti-PA IgG response reaches a threshold. The lower limit of quantification (LLOQ) is 58, results below the LLOQ have been replaced by LLOQ (58) before calculating the fold response. Thus the lowest titer that can achieve 4-fold rise is 4*58 = 232.
Time Frame: 4 weeks after the m1, m6 and m42 injections
Measure: Number (95% Confidence Interval); unit: % of participants with ≥4-fold rise
Arm/Group | Anthrax Vaccine Adsorbed 8-SQ | Anthrax Vaccine Adsorbed 8-IM | Anthrax Vaccine Adsorbed 7-IM | Anthrax Vaccine Adsorbed 5-IM | Anthrax Vaccine Adsorbed 4-IM | Anthrax Vaccine Adsorbed 754-IM | Saline Placebo IM or SQ
Number analyzed (Participants) | 235 | 234 | 139 | 141 | 157 | 698 | 243
% of participants with ≥4-fold rise
  Month 2 | 94.9 [91.3 to 97.3] | 91.9 [87.6 to 95.0] | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | 78.8 [75.6 to 81.8] | 0.4 [0.01 to 2.3]
  Month 7 | 98.6 [96.1 to 99.7] | 98.6 [96.0 to 99.7] | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | 97.8 [96.3 to 99.0] | 0.5 [0.0 to 2.5]
  Month 43 | 100.0 [97.5 to 100] | 100.0 [97.7 to 100.0] | 100.0 [97.4 to 100.0] | 99.3 [96.1 to 100.0] | 99.4 [96.5 to 100.0] | NA [NA to NA] — The 7-IM, 5-IM, and 4-IM arms received the same priming schedule, so were combined for analysis at months 2 and 7. The 754-IM arm contains the combined analysis results (months 2 and 7), the individual arms contain the month 43 results. | 0.0 [0.0 to 2.6]

ADVERSE EVENTS:
Time Frame: The observation period for Solicited AEs and Other AEs was 14 days post-injection for the first two injections, and 28 days for all subsequent injections. Serious Adverse Event (SAE) data were collected and reported to FDA as they occurred.
Description: Adverse Event data were collected for each injection during scheduled office visits and by patient reporting via a diary.
Groups:
- 8-SQ: 8 AVA injections administered subcutaneously at months 0, 0.5, 1, 6, 12, 18, 30, and 42 (the initially licensed schedule and route)
- 8-IM: 8 AVA injections administered intramuscularly at months 0, 0.5, 1, 6, 12, 18, 30, and 42
- 7-IM: 7 AVA injections administered intramuscularly at months 0, 1, 6, 12, 18, 30, and 42
- 5-IM AVA: 5 AVA injections administered intramuscularly at months 0, 1, 6, 18, and 42
- 4-IM: 4 AVA injections administered intramuscularly at months 0, 1, 6, and 42
- Saline Placebo: 8 saline placebo injections administered subcutaneously or intramuscularly at months 0, 0.5, 1, 6, 12, 18, 30, and 42. Placebo participants were grouped for analysis regardless of injection route
Arm/Group | 8-SQ | 8-IM | 7-IM | 5-IM AVA | 4-IM | Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/259 | 3/262 | 2/256 | 1/258 | 0/268 | 1/260
Serious Adverse Events (participants affected / at risk) | 26/259 | 35/262 | 27/256 | 35/258 | 38/268 | 27/260
Other Adverse Events (participants affected / at risk) | 254/259 | 250/262 | 249/256 | 253/258 | 263/268 | 200/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8-SQ (N=259) | 8-IM (N=262) | 7-IM (N=256) | 5-IM AVA (N=258) | 4-IM (N=268) | Saline Placebo (N=260)
Death due to atherosclerosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
muscle, tendon, or ligament tear/rupture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) — Due to falls, accidents, or non-specified reasons
Generalized allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Generalized allergic reaction (note: Contac Nighttime medicine was also temporally associated with some of the allergic symptoms. These symptoms reoccurred following a second exposure to Contac Nighttime medicine)
Bilateral pseudotumor cerebri (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — occurred with bilateral disc edema
Hydrocephalus and aqueductal stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — new onset of seizure led to diagnosis of hydrocephalus
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis carinii (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — stage 1A
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Basal Cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 5 (10) | 5 (5)
pancreatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
cellulitis, hospitalized (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Embolization secondary to AV malformation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prostate Cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
burns (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — following a fire
appendectomy secondary to appendicitis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Systemic Lupus Erythematosus/positive ANA (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — and lupus related disease
Traumatic Brain Injury (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — secondary to accidents (MVA, bicycle)
miscarriage/spontaneous abortion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 0 (0)
pyelonephritis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ceasarian section with healthy infant delivery (Surgical and medical procedures) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
surgical repair of cystocele, vaginocele, rectocele (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
premature labor; delivery of healthy infant (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney Stone(s) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
bypass surgery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chronic Hepatitis B (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
meningitis (viral) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acoustic Neuroma (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hospitalized for alcohol dependence/rehabilitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Angioplasty and stent placement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
staph infection secondary to poison ivy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
anemia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — secondary to fibroids and benign ovarian cyst
Thyroidectomy secondary to thyroid papillary carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
bone fracture(s) following accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) — motor vehicle, bicycle, boat
injury after falling (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — fracture or soft tissue
acute psychosis and schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
bacterial endocarditis (Cardiac disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — bacterial endocarditis (Enterococcus); persistent; weight loss and skin rash secondary to condition; led to cardiac failure and surgery (listed under "surgical procedures")
benign ovarian teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
lumbar diskectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — secondary to bilateral lumbar radiculopathy
Hospitalized for mental disorder (Psychiatric disorders) | 3 (3) | 4 (5) | 1 (1) | 0 (0) | 1 (1) | 4 (4) — to include bipolar disorder, psychosis, anxiety, depression, suicidal ideations
blood clot (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
breast reduction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
cardiac catheritization (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
head injury following motor vehicle accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — to include concussion and brain injury/coma
hospitalized for drug overdose (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
corneal ulcer/iritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
c-section; delivery of infant with bilateral congenital hip dysplasia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-section; infant with hydrocephalus and jaundice (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
c-section; infant with jaundice (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
death secondary to AIDS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
death due to suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
death due to gunshot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
death due to aneurnysm rupture (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
death due to fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
death following motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — head injury
deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dehydration secondary to other cause (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
delivery of infant with right club foot deformity (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
delivery of healthy twins (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — one vaginal, one via C-section
diverticulitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
abdominoplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
esophageal tear (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Esophageal-gastro-duodenoscopy to repair
erosive esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GI ulcers and bleeding (Gastrointestinal disorders) | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ventral hernia and repair (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hypothyroid following radioactive idodine treatment for Graves' disease (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
syncope with hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hysterectomy and salpingooophorectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
laminectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
atrial Fibrillation secondary to Mitral Valve Stenosis (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hospitalized; non-specific symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Partial paralysis following gunshot wound to head (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic Inflammatory Disease (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pituitary mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
possible C.difficile (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
possible multiple sclerosis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
post surgical complications (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — to include infection, pain at site, nausea/vomiting/constipation
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laparoscopic Lyses of Adhesions due to intestinal obstructions (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
retinal tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
intrarenal malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
shoulder impingement and correction (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
sinus reconstruction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
spleen laceration following motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stage IV Non Hodgkins Lymphoma, B cell intermediate grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
cardioconversion to correct atrial flutter with supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uncontrolled Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
uncontrolled diabetes and syncope (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
uterine fibroids (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
cholecystectomy (Surgical and medical procedures) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Lumpectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — secondary to breast cancer
metastasis of pancreatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hemicolectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — for colon cancer
pacemaker implatation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
pancreatectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
lumpectomy/mastectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
cellulitis, not hospitalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
panniculectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
mitral valve replacement (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
aortic valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
removal of vegetations due to endocarditis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — 2:1
dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) — to include heavy menses and pelvic pain
vertebral fusion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — cervical or lumbar
avascular necrosis of hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — secondary to chemotherapy and steroids
hip arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — due to avascular necrosis
prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — to remove prostate cancer
gastroesophageal reflux leading to abnormal EKG and chest pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
urosepsis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HIV positive (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
hospitalized; chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hospitalized, back pain evaluation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — no diagnosis provided
ventriculostomy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — for aqueductal stenosis
transient ischemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
benign ovarian cysts (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leiomyomata (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hysterectomy plus oophorectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
multiple injuries following motor vehicle accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — to include fractures, coma, and cardiac arrest. Patient ultimately survived injuries
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 8-SQ (N=259) | 8-IM (N=262) | 7-IM (N=256) | 5-IM AVA (N=258) | 4-IM (N=268) | Saline Placebo (N=260)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 8 | 4 | 6 | 16 | 7 | 5
ABDOMINAL PAIN NOS (Gastrointestinal disorders) | 9 | 8 | 8 | 6 | 18 | 4
DIARRHOEA NOS (Gastrointestinal disorders) | 27 | 25 | 20 | 21 | 23 | 20
DYSPEPSIA (Gastrointestinal disorders) | 16 | 12 | 16 | 13 | 25 | 21
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 13 | 8 | 8 | 9 | 12 | 13
NAUSEA (Gastrointestinal disorders) | 31 | 26 | 22 | 25 | 36 | 26
TOOTHACHE (Gastrointestinal disorders) | 14 | 16 | 11 | 8 | 11 | 11
VOMITING NOS (Gastrointestinal disorders) | 13 | 16 | 12 | 7 | 8 | 10
FATIGUE (General disorders) | 199 | 187 | 187 | 177 | 181 | 158
INJECTION SITE BRUISING (General disorders) | 150 | 101 | 85 | 101 | 80 | 74
INJECTION SITE ERYTHEMA (General disorders) | 244 | 209 | 207 | 187 | 195 | 137
INJECTION SITE JOINT MOVEMENT IMPAIRMENT (General disorders) | 163 | 179 | 177 | 176 | 188 | 42
INJECTION SITE PAIN (General disorders) | 226 | 223 | 224 | 221 | 222 | 84
INJECTION SITE PRURITUS (General disorders) | 186 | 114 | 101 | 71 | 73 | 32
INJECTION SITE SWELLING / LUMP (General disorders) | 248 | 215 | 218 | 200 | 184 | 120
INJECTION SITE TENDERNESS (General disorders) | 251 | 241 | 243 | 237 | 244 | 110
INJECTION SITE WARMTH (General disorders) | 223 | 154 | 140 | 122 | 106 | 36
PYREXIA (General disorders) | 38 | 29 | 21 | 26 | 21 | 25
HYPERSENSITIVITY NOS (Immune system disorders) | 11 | 14 | 13 | 14 | 7 | 9
INFLUENZA (Infections and infestations) | 14 | 9 | 9 | 14 | 14 | 17
NASOPHARYNGITIS (Infections and infestations) | 64 | 61 | 58 | 59 | 62 | 56
SINUSITIS NOS (Infections and infestations) | 33 | 36 | 25 | 30 | 34 | 22
UPPER RESPIRATORY TRACT INFECTION NOS (Infections and infestations) | 31 | 23 | 32 | 24 | 25 | 19
URINARY TRACT INFECTION NOS (Infections and infestations) | 9 | 19 | 15 | 9 | 8 | 23
JOINT SPRAIN (Injury, poisoning and procedural complications) | 14 | 5 | 12 | 9 | 7 | 12
LIMB INJURY NOS (Injury, poisoning and procedural complications) | 11 | 19 | 13 | 12 | 12 | 12
POST PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 22 | 18 | 15 | 13 | 21 | 21
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 11 | 17 | 9 | 12 | 6 | 13
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 57 | 50 | 45 | 50 | 52 | 44
BACK PAIN (Musculoskeletal and connective tissue disorders) | 43 | 46 | 42 | 43 | 51 | 38
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 9 | 3 | 5 | 14 | 8 | 5
MYALGIA (Musculoskeletal and connective tissue disorders) | 197 | 185 | 188 | 186 | 195 | 130
NECK PAIN (Musculoskeletal and connective tissue disorders) | 16 | 14 | 11 | 20 | 19 | 10
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 19 | 26 | 27 | 24 | 28 | 19
DIZZINESS (Nervous system disorders) | 17 | 11 | 5 | 10 | 14 | 8
HEADACHE (Nervous system disorders) | 203 | 173 | 194 | 181 | 187 | 177
ANXIETY (Psychiatric disorders) | 8 | 7 | 7 | 5 | 14 | 7
DEPRESSION (Psychiatric disorders) | 18 | 10 | 17 | 14 | 15 | 12
INSOMNIA (Psychiatric disorders) | 11 | 23 | 18 | 14 | 15 | 12
DYSMENORRHOEA (Reproductive system and breast disorders) | 22 | 21 | 27 | 17 | 30 | 25
BRONCHITIS NOS (Respiratory, thoracic and mediastinal disorders) | 17 | 10 | 16 | 18 | 16 | 7
COUGH (Respiratory, thoracic and mediastinal disorders) | 32 | 26 | 28 | 31 | 35 | 27
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 25 | 20 | 16 | 28 | 19 | 19
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 53 | 47 | 32 | 53 | 47 | 37
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 12 | 5 | 13 | 13
RHINITIS NOS (Respiratory, thoracic and mediastinal disorders) | 13 | 20 | 11 | 13 | 15 | 14
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 19 | 11 | 14 | 23 | 21 | 19
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 8 | 13 | 10 | 7 | 14 | 11
PRURITUS (Skin and subcutaneous tissue disorders) | 13 | 5 | 5 | 10 | 8 | 5
RASH NOS (Skin and subcutaneous tissue disorders) | 18 | 12 | 12 | 6 | 14 | 6
HYPERTENSION NOS (Vascular disorders) | 14 | 19 | 13 | 19 | 16 | 16

LIMITATIONS AND CAVEATS:
The study was not statistically powered to identify very rare SAEs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs must have the approval of all 5 PIs to conduct and publish additional research using clinical trial data or specimens